CLINICAL TRIAL: NCT02229227
Title: Study 200977: Albiglutide + Insulin Glargine Versus Insulin Lispro + Insulin Glargine in the Treatment of Subjects With Type 2 Diabetes Mellitus: The Switch Study
Brief Title: Safety and Efficacy of Albiglutide + Insulin Glargine Versus Insulin Lispro + Insulin Glargine Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200977; 2014-001821-34 (EudraCT Number)
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Results first posted 2018-06-29 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: switch study; albiglutide; glucagon-like peptide-1 receptor agonist; Type 2 diabetes mellitus; basal-bolus insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rGLP-1 protein; Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albiglutide + Insulin Glargine Arm (Experimental): During standardization period, subjects will transit from basal bolus regimen received during screening period to insulin glargine plus insulin lispro. During treatment period, subject will receive Albiglutide 30 milligrams (mg) weekly subcutaneous (SC) injection and insulin lispro dose will be downtitrated to half that used in the standardization period. At Week 4, Albiglutide will be uptitrated to 50 mg weekly SC injection and insulin lispro will be stopped for the remainder of the treatment Period. Insulin lispro may be re-introduced after Week 8 according to pre-defined hyperglycemia thresholds. Insulin will be adjusted according to protocol-defined insulin titration algorithms
  Interventions: Drug: Albiglutide
- Insulin Glargine + Insulin Lispro Arm (Experimental): During standardization period, subjects will transit from basal bolus regimen received during screening period to insulin glargine plus insulin lispro. During treatment period, subject will continue with the same doses as at the end of the standardization period and doses will be adjusted according to protocol-defined insulin titration algorithms
  Interventions: Drug: Insulin Glargine and Insulin Lispro

INTERVENTIONS:
Drug: Albiglutide — Albiglutide is intended for self-administration as a SC injection. It is provided as a fixed dose of 30 mg of albiglutide or 50 mg of albiglutide in a 0.5 mL injection volume, fully disposable pen injector
  Arms: Albiglutide + Insulin Glargine Arm
Drug: Insulin Glargine and Insulin Lispro — Insulin glargine and insulin lispro will be provided as injection pens for SC injection
  Arms: Insulin Glargine + Insulin Lispro Arm

SUMMARY:
This Phase IIIb, randomized, open-label, parallel group, active control, multicenter, treat to-target study of 26 weeks' treatment duration will evaluate the efficacy and safety of once-weekly albiglutide as replacement of prandial insulin in subjects with type 2 diabetes mellitus (T2DM) failing to achieve adequate glycemic control on their current basal bolus insulin regimen (with or without metformin). Approximately 794 subjects will be randomly assigned in a 1:1 ratio to 1 of 2 treatment groups: albiglutide + insulin glargine (with insulin lispro discontinuation at Week 4) (with or without metformin) or to intensification of insulin glargine + insulin lispro (with or without metformin). The study will comprise 4 study periods : Screening (2 weeks), Standardization (4 weeks), Treatment (26 weeks), and Post treatment Follow up (4 weeks). The total duration of a subject's participation will be approximately 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older (inclusive at the time of Screening) with T2DM
* HbA1c >= 7.0% and <= 9.0% at Screening.
* Currently treated with a basal-bolus insulin regimen (with or without metformin) for at least 3 months before Screening. The subject must be taking the following:
* Basal insulin (1 or 2 daily injections of neutral protamine Hagedorn insulin, insulin glargine, insulin detemir, or insulin degludec) AND
* Bolus insulin (at least 2 injections of regular insulin, insulin glulisine, insulin aspart, or insulin lispro) with a total daily dose of bolus insulin <= 70 units
* In addition, the total daily dose of insulin must be <= 140 units
* If taking metformin, a stable dose for at least 8 weeks before Screening Note: Subject should not have received any other antidiabetic medication within 30 days before screening (e.g., glucagon-like peptide-1 receptor (GLP-1R) agonist, dipeptidyl peptidase-IV inhibitor, SU, or thiazolidinedione). Subjects receiving commercially available premixed basal and prandial insulin are not eligible for this study.
* Fasting C-peptide >= 0.8 nanogram (ng) per milliliter (mL) [>= 0.26 nanomoles per litre (nmol/L)]
* Body mass index <= 40 kilogram per square meter( kg/m^2)
* Thyroid-stimulating hormone (TSH) level is normal or clinically euthyroid as demonstrated by further thyroid tests (e.g., free T4)
* Female subjects of childbearing potential (i.e., not surgically sterile and/or not postmenopausal) must be practicing adequate contraception (as defined in the protocol) for the duration of participation in the study including the 4-week post treatment Follow-up Period..
* Willing and able to comply with all study procedures including performance of frequent self-monitored blood glucose (SMBG) profiles according to the protocol
* Able and willing to provide written informed consent

Exclusion Criteria:

* Type 1 diabetes mellitus
* History of cancer that has not been in full remission for at least 3 years before Screening. (A history of squamous cell or basal cell carcinoma of the skin or treated cervical intra-epithelial neoplasia I or II is allowed)
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2
* Current symptomatic biliary disease or history of acute or chronic pancreatitis
* Severe gastroparesis, i.e., requiring regular therapy within 6 months before Screening
* History of significant GI surgery that in the opinion of the investigator is likely to significantly affect upper GI or pancreatic function [e.g., gastric bypass and banding, antrectomy, Roux-en-Y bypass, gastric vagotomy, small bowel resection, or surgeries thought to significantly affect upper GI function]
* History of severe hypoglycemia unawareness
* Diabetic complications (e.g., active proliferative retinopathy or severe diabetic neuropathy) or any other clinically significant abnormality (including a psychiatric disorder) that, in the opinion of the investigator, may pose additional risk in administering the investigational product
* Clinically significant CV and/or cerebrovascular disease within 3 months before Screening including, but not limited to, the following:
* Stroke or transient ischemic attack
* Acute coronary syndrome (myocardial infarction [MI] or unstable angina not responsive to nitroglycerin)
* Cardiac surgery or percutaneous coronary procedure
* Current or history of heart failure (New York Heart Association class III or IV)
* Alanine aminotransferase (ALT) >2.5 × upper limit of normal (ULN) or bilirubin >1.5 × ULN (isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). (Chronic stable hepatitis B and C are acceptable if subject otherwise meets entry criteria and is not on active antiviral treatment [e.g., presence of hepatitis B surface antigen or positive hepatitis C test result within 3 months of Screening])
* Hemoglobin <11 gram (g) per (dL) [<110 g/L] for male subjects and <10 g/dL (<100 g/L) for female subjects at Screening
* Estimated glomerular filtration rate (eGFR) <= 30 millilitre per minute per 1.73 square meters (mL/min/1.73 m^2) (calculated using the Modification of Diet in Renal Disease [MDRD] formula) at Screening Note: As the use of metformin in subjects with varying degrees of renal function may differ from country to country, use of metformin should be in accordance with the metformin product label within the participating country.
* Fasting triglyceride level >750 mg/dL at Screening
* Hemoglobinopathy that may affect proper interpretation of HbA1c
* Known allergy to albiglutide or any product components (including yeast and human albumin), any other GLP-1 analogue, insulin, or other study medication's excipients OR other contraindications (per the prescribing information) for the use of potential study medications (e.g., insulin glargine, insulin lispro)
* Use of oral or systemically injected glucocorticoids within the 3 months before randomization or high likelihood of a requirement for prolonged treatment (>1 week) in the 6 months following randomization. However, short courses of oral steroids (single dose or multiple doses for up to 7 days) may be permitted provided these cases are discussed with the medical monitor. Inhaled, intra-articular, epidural, and topical corticosteroids are allowed
* Female subject is pregnant (confirmed by laboratory testing) or lactating
* Receipt of any investigational drug within the 30 days or 5 half-lives, whichever is longer, before Screening, a history of receipt of an investigational antidiabetic drug within the 3 months before randomization, or receipt of albiglutide in previous studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 814 (Actual)
Dates: Start 2014-11-21 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (139):
- United States (37):
  - GSK Investigational Site, Searcy, Arkansas
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Tustin, California
  - GSK Investigational Site, West Hills, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Brooksville, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Paducah, Kentucky
  - GSK Investigational Site, Lake Charles, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Staten Island, New York
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Pharr, Texas
  - GSK Investigational Site, Round Rock, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Renton, Washington
  - GSK Investigational Site, Tacoma, Washington
- Brazil (9):
  - GSK Investigational Site, Fortaleza, Ceará
  - GSK Investigational Site, Fortaleza - CE, Ceará
  - GSK Investigational Site, Goiânia, Goiás
  - GSK Investigational Site, Uberlândia, Minas Gerais
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Campinas, São Paulo
  - GSK Investigational Site, Marília, São Paulo
  - GSK Investigational Site, Pará
  - GSK Investigational Site, São Paulo
- Canada (6):
  - GSK Investigational Site, Penticton, British Columbia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Oakville, Ontario
  - GSK Investigational Site, Thornhill, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Saint-Laurent, Quebec
- France (5):
  - GSK Investigational Site, Corbeil-Essonnes
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Valenciennes
  - GSK Investigational Site, Vandœuvre-lès-Nancy
  - GSK Investigational Site, Vénissieux
- Germany (15):
  - GSK Investigational Site, Bad Mergentheim, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Wangen, Baden-Wurttemberg
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Sulzbach-Rosenberg, Bavaria
  - GSK Investigational Site, Aßlar, Hesse
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Saarlouis, Saarland
  - GSK Investigational Site, Sankt Ingbert, Saarland
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Pirna, Saxony
  - GSK Investigational Site, Berlin
- Hungary (7):
  - GSK Investigational Site, Baja
  - GSK Investigational Site, Balatonfüred
  - GSK Investigational Site, Budaörs
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Zalaegerszeg
- Italy (5):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
- Mexico (12):
  - GSK Investigational Site, Pachuca, Hidalgo
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Monterrey NL, Nuevo León
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, Aguascalientes
  - GSK Investigational Site, Chihuahua City
  - GSK Investigational Site, Durango
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México
  - GSK Investigational Site, Veracruz
- Philippines (4):
  - GSK Investigational Site, Davao City
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Marikina City
  - GSK Investigational Site, Quezon City
- Poland (8):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Kamieniec Ząbkowicki
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Oświęcim
  - GSK Investigational Site, Puławy
  - GSK Investigational Site, Radom
  - GSK Investigational Site, Ruda Śląska
  - GSK Investigational Site, Zamość
- South Africa (6):
  - GSK Investigational Site, Bloemfontein, Free State
  - GSK Investigational Site, Johannesburg, Gauteng
  - GSK Investigational Site, Durban, KwaZulu-Natal
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Krugersdorp
  - GSK Investigational Site, Worcester
- South Korea (2):
  - GSK Investigational Site, Gyeonggido
  - GSK Investigational Site, Seoul
- Spain (18):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Alcalá de Henares
  - GSK Investigational Site, Alzira/Valencia
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barakaldo (Vizcaya)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Ferrol. La Coruña
  - GSK Investigational Site, Granada
  - GSK Investigational Site, León
  - GSK Investigational Site, Lleida
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Mérida
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia
- United Kingdom (5):
  - GSK Investigational Site, Welwyn Garden City, Hertfordshire
  - GSK Investigational Site, Bath, Somerset
  - GSK Investigational Site, Hull
  - GSK Investigational Site, Lancashire
  - GSK Investigational Site, Sidcup

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20722

REFERENCES:
- [Background] Rosenstock J, Nino A, Soffer J, Erskine L, Acusta A, Dole J, Carr MC, Mallory J, Home P. Impact of a Weekly Glucagon-Like Peptide 1 Receptor Agonist, Albiglutide, on Glycemic Control and on Reducing Prandial Insulin Use in Type 2 Diabetes Inadequately Controlled on Multiple Insulin Therapy: A Randomized Trial. Diabetes Care. 2020 Oct;43(10):2509-2518. doi: 10.2337/dc19-2316. Epub 2020 Jul 21. PMID 32694215

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 21-Nov-2014 to 24-Jul-2017 at 186 centers in 14 countries: Canada, United States of America, Mexico, Brazil, Hungary, Poland, France, Germany, Italy, Spain, United Kingdom, Korea, Philippines and South Africa.
Pre-assignment Details: A total of 2004 participants were screened, of which 973 participants were screen failures and 160 participants were re-screened. A total of 1031 participants then entered the standardization period, of which 217 participants were standardization failures. A total of 814 participants were randomized in the study.
Groups:
- Albiglutide + Insulin Glargine: During standardization period, participants transitioned from basal bolus regimen received during screening period to insulin glargine plus insulin lispro. Eligible participants received Albiglutide 30 milligrams (mg) weekly subcutaneous (SC) injection during the treatment period and insulin lispro dose was down-titrated to half that used in the standardization period. At Week 4, Albiglutide was up-titrated to 50 mg weekly SC injection and insulin lispro was stopped for the remainder of the treatment period.
- Insulin Lispro + Insulin Glargine: During standardization period, participants transitioned from basal bolus regimen received during screening period to insulin glargine plus insulin lispro. Eligible participants continued with the same doses as at the end of the standardization period and doses were adjusted according to protocol-defined insulin titration algorithms. Participants received Insulin Glargine along with Insulin Lispro during the treatment period.
Period: Overall Study
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Started | 402 | 412
Completed | 351 | 350
Not Completed | 51 | 62
Not completed — Adverse Event | 14 | 9
Not completed — Lack of Efficacy | 3 | 3
Not completed — Protocol Violation | 6 | 8
Not completed — Protocol defined stopping criteria | 1 | 3
Not completed — Lost to Follow-up | 3 | 3
Not completed — Study terminated by sponsor | 11 | 11
Not completed — Withdrawal by Subject | 8 | 12
Not completed — Other | 0 | 1
Not completed — Physician Decision | 5 | 12

BASELINE CHARACTERISTICS:
Population: Full Analysis (FA) Population comprised of all participants who were randomly assigned to treatment (who did not receive any study treatment were also included).
Groups:
- Albiglutide + Insulin Glargine: During standardization period, participants transitioned from basal bolus regimen received during screening period to insulin glargine plus insulin lispro. Eligible participants received Albiglutide 30 mg weekly SC injection during the treatment period and insulin lispro dose was down-titrated to half that used in the standardization period. At Week 4, Albiglutide was up-titrated to 50 mg weekly SC injection and insulin lispro was stopped for the remainder of the treatment period.
- Total: Total of all reporting groups
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine | Total
Number analyzed (Participants) | 402 | 412 | 814
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (9.40) | 58.1 (9.49) | 58.1 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 228 | 214 | 442
  Male | 174 | 198 | 372
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 43 | 28 | 71
  Asian-Central/South Asian (A) Heritage (H) | 5 | 8 | 13
  Asian-Japanese H/East AH/South East AH | 25 | 24 | 49
  Black or African American | 37 | 32 | 69
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  White | 284 | 312 | 596
  Multiple-Black or African American and White | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 26
Description: HbA1c is glycosylated hemoglobin. It was measured at Baseline and at Week 26. The analysis was conducted using mixed-effect model with repeated measures (MMRM). The model included HbA1c change from Baseline as the dependent variable; treatment, region, age category, current metformin use, visit week, treatment-by-week interaction, and Baseline HbA1c-by-week interaction as fixed effects; Baseline HbA1c as a continuous covariate; and participant as a random effect. The Baseline value was the last available non-missing value prior to the first dose of the randomized treatment, thus Baseline was Day -1. Change from Baseline is defined as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Day -1) and Week 26
Population: FA Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of glycosylated hemoglobin
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 345 | 350
Percentage of glycosylated hemoglobin | -1.04 (0.041) | -1.10 (0.040)
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Test type: Non-Inferiority — If the upper bound of the confidence interval is less than or equal to 0.3%, non-inferiority will be concluded; p < 0.0001, t-test, 2 sided — Non-inferiority p-value. P-value from testing the null hypothesis that the difference in change from baseline least squares means (albiglutide-insulin lispro) is greater than 0.30% based on one-sided t-test with 0.025 level of significance; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.05 to 0.17] — Least Square mean of albiglutide + insulin glargine from insulin lispro + insulin glargine has been presented

2. Secondary Outcome: Number of Participants Treated With Once-weekly Albiglutide That Were Able to Discontinue Insulin Lispro at Week 4 and Did Not Meet Prespecified Criteria for Severe, Persistent Hyperglycemia Through Week 26
Description: Participants who did not meet prespecified criteria for severe, persistent hyperglycemia through Week 26 were those participants treated with once-weekly albiglutide that were able to replace prandial insulin without lispro re-introduction through Week 26. Number of participants treated with once-weekly albiglutide that were able to discontinue insulin lispro at Week 4 and did not meet prespecified criteria for severe, persistent hyperglycemia through Week 26 have been presented.
Time Frame: Up to Week 26
Population: FA Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine
Number analyzed (Participants) | 402
Participants | 218

3. Secondary Outcome: Percentage of Participants With Severe or Documented Symptomatic Hypoglycemia Through Week 26
Description: Severe hypoglycemia was considered as an event requiring assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions. Plasma glucose concentrations may not be available during an event, but neurological recovery following the return of plasma glucose to normal was considered sufficient evidence that the event was induced by a low plasma glucose concentration. Documented symptomatic hypoglycemia was an event during which typical symptoms of hypoglycemia are accompanied by a measured plasma glucose concentration <=70 milligrams per deciliters (mg/dL) (<=3.9 millimoles per liters [mmol/L]).
Time Frame: Up to Week 26
Population: FA Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 402 | 412
Percentage of participants | 57.2 | 75.0
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — Analysis was performed using non-parametric Cochran-Mantel-Haenszel (CMH) test after adjusting for Baseline HbA1c category, age category, region and current use of metformin; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.31 to 0.60] — Odds ratio (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented

4. Secondary Outcome: Change From Baseline in Body Weight at Week 26
Description: Body weight was measured to the nearest 0.1 kilogram on a standard calibrated scale. Participants dressed in light indoor clothes (no coat, jacket, etc.) without shoes and with a voided bladder. The same equipment was used wherever possible. The Baseline value was the last available non-missing value prior to the first dose of the randomized treatment, thus Baseline was Day -1. Change from Baseline is defined as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Day -1) and Week 26
Population: FA Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Kilograms
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 349 | 352
Kilograms | -1.95 (0.207) | 2.43 (0.205)
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Test type: Superiority; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = -4.37, 95% CI 2-sided [-4.93 to -3.82] — Least Square mean difference (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented

5. Secondary Outcome: Change From Baseline to Week 26 in Body Weight
Description: Body weight was measured to the nearest 0.1 kilogram on a standard calibrated scale. Participants dressed in light indoor clothes (no coat, jacket, etc.) without shoes and with a voided bladder. The same equipment was used wherever possible. The Baseline value was the last available non-missing value prior to the first dose of the randomized treatment, thus Baseline was Day -1. Change from Baseline is defined as the post-Baseline value minus the Baseline value. Change from Baseline to Week 26 in body weight are presented. FA Population was analyzed. Only those participants available at the specified time points were analyzed represented by n=X,X in the category titles.
Time Frame: Baseline (Day -1) to Week 26
Population: FA Population.
Measure: Least Squares Mean (Standard Error); unit: Kilograms
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 402 | 412
Kilograms
  Week 4, n=368,384: number analyzed (Participants) | 368 | 384
  Week 4, n=368,384 | -0.55 (0.091) | 0.66 (0.091)
  Week 5, n=382,393: number analyzed (Participants) | 382 | 393
  Week 5, n=382,393 | -0.95 (0.102) | 0.85 (0.102)
  Week 10, n=379,397: number analyzed (Participants) | 379 | 397
  Week 10, n=379,397 | -1.71 (0.133) | 1.46 (0.131)
  Week 18, n=365,372: number analyzed (Participants) | 365 | 372
  Week 18, n=365,372 | -1.96 (0.177) | 2.06 (0.175)
  Week 26, n=349,352: number analyzed (Participants) | 349 | 352
  Week 26, n=349,352 | -1.95 (0.207) | 2.43 (0.205)
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 4; Test type: Other; Mean Difference (Net) = -1.21, 95% CI 2-sided [-1.43 to -1.00] — Least Square mean difference (albiglutide + insulin glargine minus insulin lispro + insulin glargine) at Week 4 has been presented
Statistical Analysis 2: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 5; Test type: Other; Mean Difference (Net) = -1.80, 95% CI 2-sided [-2.05 to -1.55] — Least Square mean difference (albiglutide + insulin glargine minus insulin lispro + insulin glargine) at Week 5 has been presented
Statistical Analysis 3: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 10; Test type: Other; Mean Difference (Net) = -3.17, 95% CI 2-sided [-3.51 to -2.82] — Least Square mean difference (albiglutide + insulin glargine minus insulin lispro + insulin glargine) at Week 10 has been presented
Statistical Analysis 4: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 18; Test type: Other; Mean Difference (Net) = -4.01, 95% CI 2-sided [-4.48 to -3.54] — Least Square mean difference (albiglutide + insulin glargine minus insulin lispro + insulin glargine) at Week 18 has been presented
Statistical Analysis 5: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 26; Test type: Other; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = -4.37, 95% CI 2-sided [-4.93 to -3.82] — Least Square mean difference (albiglutide + insulin glargine minus insulin lispro + insulin glargine) at Week 26 has been presented

6. Secondary Outcome: Total Daily Insulin Dose at Week 26
Description: Insulin dose at Week 26 was defined as the prescribed insulin dose at Week 25. Based on MMRM model, prescribed total daily basal insulin dose was equal to Baseline prescribed total daily basal insulin dose + treatment + Baseline HbA1c category + region + age category + current use of metformin + visit week + treatment-by-visit week interaction + Baseline prescribed total daily basal insulin dose-by-visit week interaction. Total daily insulin dose at Week 26 is presented. Only those participants available at the specified time points were analyzed.
Time Frame: Week 26
Population: FA Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: International Units
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 342 | 341
International Units | 70.36 (2.160) | 131.19 (2.149)
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Test type: Superiority; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -60.83, 95% CI 2-sided [-66.57 to -55.10] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Change From Baseline to Week 26 in HbA1c
Description: HbA1c is glycosylated hemoglobin and was measured up to Week 26. The Baseline value was the last available non-missing value prior to the first dose of the randomized treatment, thus Baseline was Day -1. Change from Baseline is defined as the post-Baseline value minus the Baseline value. Only those participants available at the specified time points were analyzed represented by n=X,X in the category titles.
Time Frame: Baseline to Week 26
Population: FA Population.
Measure: Least Squares Mean (Standard Error); unit: Percentage of glycosylated hemoglobin
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 402 | 412
Percentage of glycosylated hemoglobin
  Week 4, n=358,375: number analyzed (Participants) | 358 | 375
  Week 4, n=358,375 | -0.59 (0.023) | -0.47 (0.023)
  Week 5, n=374,392: number analyzed (Participants) | 374 | 392
  Week 5, n=374,392 | -0.67 (0.026) | -0.58 (0.025)
  Week 10, n=376,390: number analyzed (Participants) | 376 | 390
  Week 10, n=376,390 | -0.88 (0.034) | -0.96 (0.033)
  Week 18, n=360,365: number analyzed (Participants) | 360 | 365
  Week 18, n=360,365 | -1.04 (0.038) | -1.14 (0.038)
  Week 26, n=345,350: number analyzed (Participants) | 345 | 350
  Week 26, n=345,350 | -1.04 (0.041) | -1.1 (0.040)
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 4; Test type: Non-Inferiority — Difference in change from Baseline least squares means (albiglutide - insulin lispro) is greater than 0.30% based on one-sided t-test with 0.025 level of significance; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.18 to -0.07] — Least square mean difference (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented for Week 4
Statistical Analysis 2: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 5; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.15 to -0.02] — Least square mean difference (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented for Week 5
Statistical Analysis 3: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 10; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.01 to 0.17] — Least square mean difference (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented for Week 10
Statistical Analysis 4: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 18; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = 0.11, 95% CI 2-sided [0.01 to 0.21] — Least square mean difference (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented for Week 18
Statistical Analysis 5: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 26; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.05 to 0.17] — Least square mean difference (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented for Week 26

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26
Description: FPG was measured at Baseline (Day -1). FPG values for all participants at Week 26 were not collected due to an error in the protocol and were imputed with the fasting serum glucose (FSG) values at this time point. The imputation of the FPG at Week 26 from the FSG values was deemed acceptable from the results of the analysis of the correlation between FPG and FSG at the screening visit. The Baseline value was the last available non-missing value prior to the first dose of the randomized treatment, thus Baseline was Day -1. Change from Baseline is defined as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 26
Population: FA Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per Liter
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 345 | 349
Millimoles per Liter | -2.01 (0.120) | -1.46 (0.121)
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Test type: Superiority; p = 0.0004, t-test, 2 sided; Mean Difference (Net) = -0.55, 95% CI 2-sided [-0.86 to -0.25] — [estimate comment as in outcome 4, analysis 1]

9. Secondary Outcome: Change From Baseline to Week 26 in FPG
Description: FPG was measured at Baseline (Day -1) up to Week 26. FPG values for all participants at Week 26 were not collected due to an error in the protocol and were imputed with the FSG values at this time point. The imputation of the FPG at Week 26 from the FSG values was deemed acceptable from the results of the analysis of the correlation between FPG and FSG at the screening visit. The Baseline value was the last available non-missing value prior to the first dose of the randomized treatment, thus Baseline was Day -1. Change from Baseline is defined as the post-Baseline value minus the Baseline value.
Time Frame: Baseline to Week 26
Population: FA Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per Liter
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 402 | 412
Millimoles per Liter
  Week 4, n=356,371: number analyzed (Participants) | 356 | 371
  Week 4, n=356,371 | -1.30 (0.119) | -0.76 (0.118)
  Week 5, n=366,388: number analyzed (Participants) | 366 | 388
  Week 5, n=366,388 | -1.07 (0.126) | -0.88 (0.125)
  Week 18, n=348,353: number analyzed (Participants) | 348 | 353
  Week 18, n=348,353 | -1.76 (0.124) | -1.23 (0.124)
  Week 26, n=345,349: number analyzed (Participants) | 345 | 349
  Week 26, n=345,349 | -2.01 (0.120) | -1.46 (0.121)
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 4; Test type: Other; Mean Difference (Net) = -0.54, 95% CI 2-sided [-0.84 to -0.24] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 5; Test type: Other; Mean Difference (Net) = -0.19, 95% CI 2-sided [-0.51 to 0.13] — [estimate comment as in outcome 7, analysis 2]
Statistical Analysis 3: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 18; Test type: Other; Mean Difference (Net) = -0.53, 95% CI 2-sided [-0.85 to -0.22] — [estimate comment as in outcome 7, analysis 4]
Statistical Analysis 4: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 26; Test type: Superiority; p = 0.0004, t-test, 2 sided; Mean Difference (Net) = -0.55, 95% CI 2-sided [-0.86 to -0.25] — [estimate comment as in outcome 7, analysis 5]

10. Secondary Outcome: Number of Participants Achieving HbA1c <7.0% at Week 26
Description: HbA1c is glycosylated hemoglobin. Number of participants achieving a HbA1c <7.0% at Week 26 are presented.
Time Frame: Week 26
Population: FA Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 402 | 412
Participants | 244 | 255
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Test type: Other; p = 0.7026, Cochran-Mantel-Haenszel — Non-parametric Cochran-Mantel-Haenszel (CMH) test after adjusting for Baseline HbA1c category, age category, region and current use of metformin; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.71 to 1.31] — Odds ratio (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented

11. Secondary Outcome: Number of Participants Achieving HbA1c <7.0% up to Week 26
Description: HbA1c is glycosylated hemoglobin. Number of participants achieving a HbA1c <7.0% up to Week 26 are presented.
Time Frame: Up to Week 26
Population: FA Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 402 | 412
Participants
  Week 4 | 142 | 139
  Week 5 | 157 | 182
  Week 10 | 220 | 261
  Week 18 | 251 | 281
  Week 26 | 244 | 255
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 4; Test type: Other; p = 0.2883, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.84 to 1.64] — Odds ratio (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented for Week 4
Statistical Analysis 2: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 5; Test type: Other; p = 0.3034, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.59 to 1.15] — Odds ratio (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented for Week 5
Statistical Analysis 3: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 10; Test type: Other; p = 0.0151, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.52 to 0.98] — Odds ratio (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented for Week 10
Statistical Analysis 4: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 18; Test type: Other; p = 0.0518, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.54 to 1.03] — Odds ratio (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented for Week 18
Statistical Analysis 5: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 26; Test type: Other; p = 0.7026, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.71 to 1.31] — Odds ratio (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented for Week 26

12. Secondary Outcome: Number of Participants Achieving a HbA1c <6.5% at Week 26
Description: Number of participants achieving a HbA1c <6.5% at Week 26 are presented.
Time Frame: Week 26
Population: FA Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 402 | 412
Participants | 147 | 169
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Test type: Other; p = 0.2298, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.63 to 1.17] — Odds ratio (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented

13. Secondary Outcome: Number of Participants Achieving a HbA1c <6.5% up to Week 26
Description: Number of participants achieving a HbA1c <6.5% up to Week 26 are presented.
Time Frame: Up to Week 26
Population: FA Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 402 | 412
Participants
  Week 4 | 39 | 33
  Week 5 | 63 | 62
  Week 10 | 116 | 140
  Week 18 | 150 | 178
  Week 26 | 147 | 169
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 4; Test type: Other; p = 0.2143, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.78 to 2.23] — Odds ratio (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented for Week 4
Statistical Analysis 2: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 5; Test type: Other; p = 0.4703, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.80 to 1.91] — Odds ratio (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented for Week 5
Statistical Analysis 3: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 10; Test type: Other; p = 0.2139, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.58 to 1.14] — Odds ratio (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented for Week 10
Statistical Analysis 4: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 18; Test type: Other; p = 0.0790, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.59 to 1.11] — Odds ratio (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented for Week 18
Statistical Analysis 5: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 26; Test type: Other; p = 0.2298, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.63 to 1.17] — Odds ratio (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented for Week 26

14. Secondary Outcome: Number of Participants Who Met Prespecified Criteria for Severe, Persistent Hyperglycemia at Week 26
Description: Meeting prespecified criteria for severe, persistent hyperglycemia was defined operationally as being withdrawn due to lack of efficacy as recorded on the Treatment Discontinuation and Study Conclusion electronic case report form pages. Number of participants who met prespecified criteria for severe, persistent hyperglycemia at Week 26 are presented.
Time Frame: Week 26
Population: FA Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 402 | 412
Participants | 3 | 3
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Test type: Other; p = 0.8292, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.24 to 4.77] — Odds ratio (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented

15. Secondary Outcome: Number of Participants Meeting Prespecified Criteria for Severe, Persistent Hyperglycemia up to Week 26
Description: Meeting prespecified criteria for severe, persistent hyperglycemia was defined operationally as being withdrawn due to lack of efficacy as recorded on the Treatment Discontinuation and Study Conclusion electronic case report form pages. Number of participants meeting prespecified criteria for severe, persistent hyperglycemia up to Week 26 are presented.
Time Frame: Up to Week 26
Population: FA Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 402 | 412
Participants
  0 to <=4 Weeks | 0 | 0
  >4 to <=5 Weeks | 0 | 0
  >5 to <=10 Weeks | 2 | 0
  >10 to <=18 Weeks | 0 | 1
  >18 to <=26 Weeks | 1 | 2

16. Secondary Outcome: Total Daily Insulin Dose at Week 4, Week 10 and Week 18
Description: Based on MMRM model, prescribed total daily basal insulin dose was equal to Baseline prescribed total daily basal insulin dose + treatment + Baseline HbA1c category + region + age category + current use of metformin + visit week + treatment-by-visit week interaction + Baseline prescribed total daily basal insulin dose-by-visit week interaction. Total daily insulin dose at Week 4, Week 10 and Week 18 is presented. Only those participants available at the specified time points were analyzed represented by n=X,X in the category titles.
Time Frame: Weeks 4, 10, and 18
Population: FA Population.
Measure: Least Squares Mean (Standard Error); unit: International Units
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 402 | 412
International Units
  Week 4, n=388,403: number analyzed (Participants) | 388 | 403
  Week 4, n=388,403 | 50.53 (1.183) | 106.91 (1.187)
  Week 10, n=375,386: number analyzed (Participants) | 375 | 386
  Week 10, n=375,386 | 57.99 (1.597) | 121.69 (1.589)
  Week 18, n=359,361: number analyzed (Participants) | 359 | 361
  Week 18, n=359,361 | 68.23 (2.010) | 130.22 (1.998)
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 4; Test type: Other; Mean Difference (Final Values) = -56.38, 95% CI 2-sided [-59.19 to -53.57] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 10; Test type: Other; Mean Difference (Final Values) = -63.70, 95% CI 2-sided [-67.78 to -59.62] — [estimate comment as in outcome 7, analysis 3]
Statistical Analysis 3: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 18; Test type: Other; Mean Difference (Final Values) = -62.00, 95% CI 2-sided [-67.29 to -56.70] — [estimate comment as in outcome 7, analysis 4]

17. Secondary Outcome: Total Daily Basal Insulin (Insulin Glargine) at Week 4, 10, 18, and 26 Visits
Description: Based on MMRM model, prescribed total daily basal insulin dose was equal to Baseline prescribed total daily basal insulin dose + treatment + Baseline HbA1c category + region + age category + current use of metformin + visit week + treatment-by-visit week interaction + Baseline prescribed total daily basal insulin dose-by-visit week interaction. Total daily basal insulin (insulin glargine) at Week 4, 10, 18, and 26 visits is presented. Only those participants available at the specified time points were analyzed represented by n=X,X in the category titles.
Time Frame: Weeks 4, 10, 18, and 26
Population: FA Population.
Measure: Least Squares Mean (Standard Error); unit: International Units
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 402 | 412
International Units
  Week 4, n=388,403: number analyzed (Participants) | 388 | 403
  Week 4, n=388,403 | 49.97 (0.534) | 50.94 (0.536)
  Week 10, n=375,386: number analyzed (Participants) | 375 | 386
  Week 10, n=375,386 | 56.14 (0.767) | 55.79 (0.761)
  Week 18, n=359,361: number analyzed (Participants) | 359 | 361
  Week 18, n=359,361 | 59.42 (0.928) | 59.18 (0.920)
  Week 26, n=342,341: number analyzed (Participants) | 342 | 341
  Week 26, n=342,341 | 59.83 (0.996) | 59.43 (0.988)
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 4; Test type: Superiority; Mean Difference (Final Values) = -0.97, 95% CI 2-sided [-2.25 to 0.30] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 10; Test type: Other; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-1.64 to 2.33] — [estimate comment as in outcome 7, analysis 3]
Statistical Analysis 3: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 18; Test type: Other; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-2.21 to 2.69] — [estimate comment as in outcome 7, analysis 4]
Statistical Analysis 4: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 26; Test type: Other; p = 0.7699, t-test, 2 sided; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [-2.25 to 3.04] — [estimate comment as in outcome 7, analysis 5]

18. Secondary Outcome: Total Daily Bolus Insulin (Insulin Lispro) at Week 4, 10, 18, and 26 Visits
Description: Based on MMRM model, prescribed total daily basal insulin dose was equal to Baseline prescribed total daily basal insulin dose + treatment + Baseline HbA1c category + region + age category + current use of metformin + visit week + treatment-by-visit week interaction + Baseline prescribed total daily basal insulin dose-by-visit week interaction. Total daily bolus insulin (insulin lispro) at Week 4, 10, 18, and 26 visits is presented. Only those participants available at the specified time points were analyzed represented by n=X,X in the category titles.
Time Frame: Weeks 4, 10, 18, and 26
Population: FA Population.
Measure: Least Squares Mean (Standard Error); unit: International Units
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 402 | 412
International Units
  Week 4, n=388,403: number analyzed (Participants) | 388 | 403
  Week 4, n=388,403 | 0.62 (0.887) | 56.67 (0.892)
  Week 10, n=375,386: number analyzed (Participants) | 375 | 386
  Week 10, n=375,386 | 1.90 (1.147) | 66.66 (1.144)
  Week 18, n=359,361: number analyzed (Participants) | 359 | 361
  Week 18, n=359,361 | 8.89 (1.436) | 71.81 (1.430)
  Week 26, n=342,341: number analyzed (Participants) | 342 | 341
  Week 26, n=342,341 | 10.64 (1.523) | 72.47 (1.517)
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 4; Test type: Other; Mean Difference (Final Values) = -56.05, 95% CI 2-sided [-58.17 to -53.94] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 10; Test type: Other; Mean Difference (Final Values) = -64.76, 95% CI 2-sided [-67.68 to -61.85] — [estimate comment as in outcome 7, analysis 3]
Statistical Analysis 3: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Week 18; Test type: Other; Mean Difference (Final Values) = -62.92, 95% CI 2-sided [-66.69 to -59.15] — [estimate comment as in outcome 7, analysis 4]
Statistical Analysis 4: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; week 26; Test type: Superiority; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -61.83, 95% CI 2-sided [-65.85 to -57.81] — [estimate comment as in outcome 7, analysis 5]

19. Secondary Outcome: Total Number of Weekly Insulin Injections to Achieve Glycemic Control at Baseline/Randomization and Week 4, 10, 18, and 26
Description: Total number of weekly insulin injections (7 days) to achieve glycemic control at Baseline/Randomization and Week 4, 10, 18, and 26 are presented. Only those participants available at the specified time points were analyzed represented by n=X,X in category titles.
Time Frame: Baseline (Day -1) and Weeks 4, 10, 18 and 26
Population: FA Population.
Measure: Mean (Standard Deviation); unit: Insulin Injections
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 402 | 412
Insulin Injections
  Baseline, n=401,412: number analyzed (Participants) | 401 | 412
  Baseline, n=401,412 | 28.79 (1.470) | 28.00 (0.000)
  Week 4, n=388,403: number analyzed (Participants) | 388 | 403
  Week 4, n=388,403 | 8.11 (1.506) | 28.00 (0.000)
  Week 10, n=375,386: number analyzed (Participants) | 375 | 386
  Week 10, n=375,386 | 9.06 (3.121) | 28.00 (0.000)
  Week 18, n=359,361: number analyzed (Participants) | 359 | 361
  Week 18, n=359,361 | 12.62 (7.330) | 28.00 (0.000)
  Week 26, n=342,341: number analyzed (Participants) | 342 | 341
  Week 26, n=342,341 | 13.22 (7.758) | 28.00 (0.000)

20. Secondary Outcome: Percentage of Participants Achieving HbA1c <7.0% Without Weight Gain at Week 26
Description: Percentage of participants achieving HbA1c <7.0% without weight gain are presented.
Time Frame: Week 26
Population: FA Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 402 | 412
Percentage of participants | 49.8 | 21.4
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 3.50, 95% CI 2-sided [2.52 to 4.86] — Odds ratio (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented

21. Secondary Outcome: Percentage of Participants Achieving HbA1c <7.0% Without Severe or Documented Symptomatic Hypoglycemia at Week 26
Description: Percentage of participants achieving HbA1c <7.0% without severe or documented symptomatic hypoglycemia are presented.
Time Frame: Week 26
Population: FA Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 402 | 412
Percentage of participants | 21.1 | 9.5
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 2.36, 95% CI 2-sided [1.54 to 3.60] — Odds ratio (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented

22. Secondary Outcome: Percentage of Participants Achieving HbA1c <7.0% Without Weight Gain and Without Severe or Documented Hypoglycemia at Week 26
Description: Percentage of participants achieving HbA1c <7.0% without weight gain and without severe or documented hypoglycemia are presented.
Time Frame: Week 26
Population: FA Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 402 | 412
Percentage of participants | 15.9 | 3.9
Statistical Analysis 1: Comparison: Albiglutide + Insulin Glargine vs Insulin Lispro + Insulin Glargine; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 3.78, 95% CI 2-sided [2.21 to 6.48] — Odds ratio (albiglutide + insulin glargine minus insulin lispro + insulin glargine) has been presented

23. Secondary Outcome: Number of Participants With On-therapy Adverse Events (AE) and Serious AE (SAE), and AE Leading to Discontinuation of Randomized Study Medication
Description: AE is any untoward medical occurrence in a participant, temporally associated with use of medicinal product (MP), whether or not considered related to MP. AE can be any unfavorable, unintended sign (also an abnormal laboratory finding), symptom, or disease (new/exacerbated) temporally associated with use of MP. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, or is a congenital anomaly/birth defect or is medically significant or all events of possible drug induced liver injury with hyperbilirubinemia. Safety Population: All participants who received at least 1 dose of randomized study medication. A participant randomized to Albiglutide + Insulin glargine by mistake received Insulin Lispro + Insulin Glargine instead. Since this participant received actual treatment as Insulin Lispro + Insulin Glargine, was summarized as such in Safety Population.
Time Frame: Up to Week 26
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 400 | 413
Participants
  AE | 261 | 254
  SAE | 23 | 31
  AE leading to study medication discontinuation | 12 | 6

24. Secondary Outcome: Number of Participants With Other AE of Special Interest
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with use of a MP, whether or not considered related to MP. AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with use of MP. AE of special interest included hypoglycemic events, cardiovascular events, gastrointestinal events, injection site reactions, potential systemic allergic reactions, pancreatitis, pancreatic cancer, malignant neoplasms following treatment with insulin, diabetic retinopathy events, appendicitis, liver events, pneumonia, and atrial fibrillation/flutter.
Time Frame: Up to Week 26
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 400 | 413
Participants
  Hypoglycemic Events | 305 | 361
  Cardiovascular Events | 7 | 9
  Gastrointestinal Events | 102 | 53
  Injection Site Reactions | 8 | 1
  Systemic Allergic Reactions | 3 | 0
  Pancreatitis | 1 | 0
  Pancreatic cancer | 0 | 0
  Malignant Neoplasm | 2 | 2
  Diabetic Retinopathy | 4 | 17
  Appendicitis | 1 | 0
  Liver Events | 0 | 2
  Pneumonia | 1 | 3
  Atrial Fibrillation/Flutter | 4 | 1

25. Secondary Outcome: Percentage of Participants With Events of Hypoglycemia With Confirmed Home Blood Glucose Monitoring and/or Third-party Intervention Through Week 26
Description: Hypoglycemic events with confirmed home plasma glucose monitoring <3.9 millimoles per Liter and/or requiring third party intervention were severe, documented symptomatic (DS) and asymptomatic hypoglycemic events. Participants with more than one hypoglycemic event are counted in all categories reported. Any severe, documented symptomatic, and asymptomatic hypoglycemic events in 3-month intervals (i.e., from Day 0 to Week 12, >Week 12 to Week 26) are presented.
Time Frame: Up to Week 26
Population: Safety Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 400 | 413
Percentage of participants
  Any event: Onset date falls under 0 to <= 12 weeks | 55.3 | 79.2
  Any event: Onset date falls > 12 to <= 26 Weeks | 60.3 | 79.4
  Severe: Onset date falls under 0 to <= 12 weeks | 1.8 | 3.6
  Severe: Onset date falls > 12 to <= 26 Weeks | 0.8 | 1.9
  DS: Onset date falls under 0 to <= 12 weeks | 33.8 | 63.0
  DS: Onset date falls > 12 to <= 26 Weeks | 40.8 | 62.0
  Asymptomatic: Onset date under 0 to <= 12 weeks | 38.3 | 56.9
  Asymptomatic: Onset date falls > 12 to <= 26 Weeks | 44.3 | 54.7

26. Secondary Outcome: Number of Participants With Hypoglycemic Events (in Total and by Each Category as Defined by the American Diabetes Association Criteria)
Description: The American Diabetes Association has categorized hypoglycemic events as follows: Severe, documented symptomatic, asymptomatic, probably symptomatic and pseudohypoglycemia. Number of participants with hypoglycemic events in total are also presented.
Time Frame: Up to Week 26
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 400 | 413
Participants
  Severe | 9 | 22
  Documented Symptomatic | 203 | 299
  Asymptomatic | 230 | 293
  Probably Symptomatic | 29 | 52
  Pseudohypoglycemia | 45 | 83
  Missing | 9 | 13
  Total | 305 | 361

27. Secondary Outcome: Number of Participants With Daytime and Nocturnal Hypoglycemia
Description: Daytime hypoglycemia was defined as hypoglycemic events with an onset between 06:00 hours and 00:00 hours (inclusive), and nocturnal hypoglycemia (in total and by category), defined as hypoglycemic events with an onset between 00:01 hours and 05:59 hours (inclusive). Number of participants with daytime and nocturnal hypoglycemia (in total and by category) are presented.
Time Frame: Up to Week 26
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 400 | 413
Participants
  Any (Total) Daytime Hypoglycemic Event | 288 | 356
  Any (Total) Nocturnal Hypoglycemic Event | 155 | 225
  Severe Daytime Hypoglycemic Event | 6 | 14
  Severe Nocturnal Hypoglycemic Event | 4 | 6
  Documented Symptomatic Daytime Hypoglycemic event | 187 | 293
  Documented Symptomatic Nocturnal Hypoglycemia | 101 | 152
  Asymptomatic Daytime Hypoglycemic event | 217 | 281
  Asymptomatic Nocturnal Hypoglycemic event | 77 | 106
  Probably Symptomatic Daytime Hypoglycemic event | 22 | 44
  Probably Symptomatic Nocturnal Hypoglycemic event | 7 | 21
  Pseudohypoglycemia Daytime Hypoglycemic event | 36 | 70
  Pseudohypoglycemia Nocturnal Hypoglycemic event | 17 | 34
  Missing Daytime Hypoglycemic Event | 9 | 11
  Mising Nocturnal Hypoglycemic Event | 2 | 4

28. Secondary Outcome: Number of Participants With Hypoglycemia With Blood Glucose <56 Milligrams Per Deciliter (mg/dL) (<3.1 Millimoles Per Liter [mmol/L]), Regardless of Symptoms
Description: Number of participants with hypoglycemia with blood glucose <56 mg/dL (<3.1 mmol/L), regardless of symptoms are presented.
Time Frame: Up to Week 26
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 400 | 413
Participants | 141 | 239

29. Secondary Outcome: Number of Participants With Hematology Values of Clinical Concern
Description: Hematology parameters included basophils, eosinophils, hematocrit, hemoglobin, lymphocytes, monocytes, neutrophils, neutrophil bands, platelets, red blood cell (RBC) count, segmented neutrophils and white blood cell (WBC) count. The potential clinical concern values were: Hematocrit >0.05 below lower limit of normal (LLN) and >0.04 above upper limit of normal (ULN), hemoglobin: >20 grams cells per Liter (g/L) below LLN and >10 g/L above ULN, lymphocytes: <0.5 x LLN, neutrophils: <1 giga cells per liter (GI/L), platelets: <80 GI/L and >500 GI/L, segmented neutrophils: <0.5 x LLN, RBC count: >1 GI/L below LLN and >5 GI/L above ULN and none for basophils, eosinophils, monocytes, neutrophil bands and RBC count. Only those parameters for which at least one value of potential clinical concern was reported are summarized.
Time Frame: Up to 30 weeks
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 394 | 407
Participants
  Hematocrit: >0.05 (fraction) below LLN | 5 | 6
  Hematocrit: >0.04 (fraction) above ULN | 9 | 12
  Hemoglobin: >20 g/L below LLN | 9 | 9
  Hemoglobin: >10 g/L above ULN | 2 | 3
  Leukocytes: >1 GI/L below LLN | 1 | 1
  Leukocytes: >5 GI/L above ULN | 4 | 1
  Neutrophils: <1 GI/L | 2 | 3
  Neutrophils, Segmented: <0.5 x LLN | 2 | 3
  Platelets: <80 GI/L | 1 | 1
  Platelets: >500 GI/L | 3 | 1

30. Secondary Outcome: Number of Participants With Clinical Chemistry Values of Clinical Concern
Description: Clinical chemistry parameters and their potential clinical concern values were: albumin (>5 g/L above ULN or below LLN), alkaline phosphatase(>3 x ULN), alanine aminotransferase (>3 x ULN), aspartate aminotransferase (>3 x ULN), carbon dioxide content (<16 millimoles per Liter [mmol/L] and > 40 mmol/L), blood urea nitrogen (>2 x ULN), calcium (<1.8 mmol/L and >3.0 mmol/L), chloride (none), creatinine (>159 micromoles/Liter), direct bilirubin (>1.35 x ULN), gamma glutamyl transferase (>3 x ULN), glucose (fasting) (<3 mmol/L and >22 mmol/L), magnesium (<0.411 mmol/L and >1.644 mmol/L), phosphate (>0.323 mmol/L above ULN or below LLN), potassium (>0.5 mmol/L below LLN and >1.0 mmol/L above ULN), sodium (>5 mmol/L above ULN or below LLN), triglycerides (> 9.04 mmol/L), total bilirubin (>1.5 x ULN), total protein (>15 g/L above ULN or below LLN) and uric acid (>654 umol/L). Only those parameters for which at least one value of potential clinical concern was reported are summarized.
Time Frame: Up to 30 weeks
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 400 | 413
Participants
  Fasting Serum Glucose: <3 mmol/L, n= 394,405: number analyzed (Participants) | 394 | 405
  Fasting Serum Glucose: <3 mmol/L, n= 394,405 | 12 | 16
  Fasting Serum Glucose: >22 mmol/L, n= 394,405: number analyzed (Participants) | 394 | 405
  Fasting Serum Glucose: >22 mmol/L, n= 394,405 | 0 | 1
  Fasting Plasma Glucose: <3 mmol/L, n= 388,406: number analyzed (Participants) | 388 | 406
  Fasting Plasma Glucose: <3 mmol/L, n= 388,406 | 9 | 14
  Fasting Plasma Glucose: >22 mmol/L, n= 388,406: number analyzed (Participants) | 388 | 406
  Fasting Plasma Glucose: >22 mmol/L, n= 388,406 | 1 | 0
  Albumin: >5 g/L below LLN, n=394,407: number analyzed (Participants) | 394 | 407
  Albumin: >5 g/L below LLN, n=394,407 | 0 | 0
  Albumin: >5 g/L above ULN, n=394,407: number analyzed (Participants) | 394 | 407
  Albumin: >5 g/L above ULN, n=394,407 | 0 | 0
  Calcium: <1.8 mmol/L, n=394,407: number analyzed (Participants) | 394 | 407
  Calcium: <1.8 mmol/L, n=394,407 | 1 | 1
  Calcium: >3.0 mmol/L, n=394,407: number analyzed (Participants) | 394 | 407
  Calcium: >3.0 mmol/L, n=394,407 | 0 | 0
  Carbon Dioxide: <16 mmol/L, n=394,407: number analyzed (Participants) | 394 | 407
  Carbon Dioxide: <16 mmol/L, n=394,407 | 5 | 8
  Carbon Dioxide: >40 mmol/L, n=394,407: number analyzed (Participants) | 394 | 407
  Carbon Dioxide: >40 mmol/L, n=394,407 | 0 | 0
  Magnesium: <0.411 mmol/L, n=394,407: number analyzed (Participants) | 394 | 407
  Magnesium: <0.411 mmol/L, n=394,407 | 1 | 1
  Magnesium: >1.644 mmol/L, n=394,407: number analyzed (Participants) | 394 | 407
  Magnesium: >1.644 mmol/L, n=394,407 | 0 | 0
  Phosphate: >0.323 mmol/L below LLN, n=394,407: number analyzed (Participants) | 394 | 407
  Phosphate: >0.323 mmol/L below LLN, n=394,407 | 0 | 0
  Phosphate: >0.323 mmol/L above ULN, n=394,407: number analyzed (Participants) | 394 | 407
  Phosphate: >0.323 mmol/L above ULN, n=394,407 | 2 | 4
  Potassium: >0.5 mmol/L below LLN, n=394,407: number analyzed (Participants) | 394 | 407
  Potassium: >0.5 mmol/L below LLN, n=394,407 | 1 | 0
  Potassium: >1.0 mmol/L above ULN, n=394,407: number analyzed (Participants) | 394 | 407
  Potassium: >1.0 mmol/L above ULN, n=394,407 | 0 | 1
  Protein: >15 g/L below LLN, n=394,407: number analyzed (Participants) | 394 | 407
  Protein: >15 g/L below LLN, n=394,407 | 0 | 0
  Protein: >15 g/L above ULN, n=394,407: number analyzed (Participants) | 394 | 407
  Protein: >15 g/L above ULN, n=394,407 | 0 | 0
  Sodium: >5 mmol/L below LLN, n=394,407: number analyzed (Participants) | 394 | 407
  Sodium: >5 mmol/L below LLN, n=394,407 | 1 | 0
  Sodium: >5 mmol/L above ULN, n=394,407: number analyzed (Participants) | 394 | 407
  Sodium: >5 mmol/L above ULN, n=394,407 | 1 | 0
  Triglycerides: >9.04 mmol/L, n=393,405: number analyzed (Participants) | 393 | 405
  Triglycerides: >9.04 mmol/L, n=393,405 | 7 | 1
  Urate: >654 μmol/L, n=394,407: number analyzed (Participants) | 394 | 407
  Urate: >654 μmol/L, n=394,407 | 0 | 2
  Urea: >2 x ULN, n=394,407: number analyzed (Participants) | 394 | 407
  Urea: >2 x ULN, n=394,407 | 2 | 1
  Alanine Aminotransferase: >3 x ULN, n=396,410: number analyzed (Participants) | 396 | 410
  Alanine Aminotransferase: >3 x ULN, n=396,410 | 0 | 5
  Alkaline Phosphatase: >3 x ULN, n=396,410: number analyzed (Participants) | 396 | 410
  Alkaline Phosphatase: >3 x ULN, n=396,410 | 1 | 0
  Aspartate Aminotransferase: >3 x ULN, n=396,410: number analyzed (Participants) | 396 | 410
  Aspartate Aminotransferase: >3 x ULN, n=396,410 | 0 | 2
  Bilirubin: >1.5 x ULN, n=396,410: number analyzed (Participants) | 396 | 410
  Bilirubin: >1.5 x ULN, n=396,410 | 1 | 1
  Creatinine: >159 μmol/L, n=396,410: number analyzed (Participants) | 396 | 410
  Creatinine: >159 μmol/L, n=396,410 | 20 | 16
  Direct Bilirubin: >1.35 x ULN, n=396,410: number analyzed (Participants) | 396 | 410
  Direct Bilirubin: >1.35 x ULN, n=396,410 | 0 | 1
  Gamma Glutamyl Transferase: >3 x ULN, n=396,410: number analyzed (Participants) | 396 | 410
  Gamma Glutamyl Transferase: >3 x ULN, n=396,410 | 14 | 14

31. Secondary Outcome: Mean Urine Albumin/Creatinine Ratio at Week 0 and Week 26
Description: Urine samples were collected for analysis of albumin/creatinine ratio. Only those participants available at the specified time points were analyzed represented by n=X,X in the category titles. Mean urine albumin/creatinine ratio at Week 0 and Week 26 are presented.
Time Frame: Week 0 and Week 26
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per mole
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 400 | 413
Grams per mole
  Week 0, n=369,376: number analyzed (Participants) | 369 | 376
  Week 0, n=369,376 | 14.40 (49.884) | 11.57 (31.089)
  Week 26, n=317,324: number analyzed (Participants) | 317 | 324
  Week 26, n=317,324 | 10.37 (32.992) | 11.55 (31.975)

32. Secondary Outcome: Mean Albumin at Week 0 and Week 26
Description: Urine samples were collected for analysis of albumin. Only those participants available at the specified time points were analyzed represented by n=X,X in the category titles. Mean albumin at Week 0 and Week 26 are presented.
Time Frame: Week 0 and Week 26
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milligrams per Liter
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 400 | 413
Milligrams per Liter
  Week 0, n=394,405: number analyzed (Participants) | 394 | 405
  Week 0, n=394,405 | 127.7 (428.46) | 108.2 (301.88)
  Week 26, n=348,345: number analyzed (Participants) | 348 | 345
  Week 26, n=348,345 | 110.5 (375.41) | 146.3 (628.73)

33. Secondary Outcome: Mean Creatinine at Week 0 and Week 26
Description: Urine samples were collected for analysis of creatinine. Only those participants available at the specified time points were analyzed represented by n=X,X in the category titles. Mean creatinine at Week 0 and Week 26 are presented.
Time Frame: Week 0 and Week 26
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per Liter
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 400 | 413
Micromoles per Liter
  Week 0, n=395,406: number analyzed (Participants) | 395 | 406
  Week 0, n=395,406 | 10646.3 (5190.43) | 10663.8 (5639.54)
  Week 26, n=350,345: number analyzed (Participants) | 350 | 345
  Week 26, n=350,345 | 11364.6 (5998.72) | 11394.2 (5663.72)

34. Secondary Outcome: Mean Specific Gravity at Week 0 and Week 26
Description: Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. A urinary specific gravity measurement is a routine part of urinalysis. Only those participants available at the specified time points were analyzed represented by n=X,X in the category titles.
Time Frame: Week 0 and Week 26
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 400 | 413
Ratio
  Week 0, n=388,402: number analyzed (Participants) | 388 | 402
  Week 0, n=388,402 | 1.0182 (0.00599) | 1.0180 (0.00588)
  Week 26, n=347,343: number analyzed (Participants) | 347 | 343
  Week 26, n=347,343 | 1.0180 (0.00627) | 1.0186 (0.00588)

35. Secondary Outcome: Number of Participants With Different Values of Potential of Hydrogen (pH) at Week 0 and Week 26
Description: Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Safety Population was analyzed. Only those participants available at the specified time points were analyzed represented by n=X,X in the category titles.
Time Frame: Week 0 and Week 26
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 400 | 413
Participants
  pH=5; Week 0, n=388,402: number analyzed (Participants) | 388 | 402
  pH=5; Week 0, n=388,402 | 92 | 107
  pH=5.5; Week 0, n=388,402: number analyzed (Participants) | 388 | 402
  pH=5.5; Week 0, n=388,402 | 132 | 132
  pH=6; Week 0, n=388,402: number analyzed (Participants) | 388 | 402
  pH=6; Week 0, n=388,402 | 86 | 77
  pH=6.5; Week 0, n=388,402: number analyzed (Participants) | 388 | 402
  pH=6.5; Week 0, n=388,402 | 29 | 43
  pH=7; Week 0, n=388,402: number analyzed (Participants) | 388 | 402
  pH=7; Week 0, n=388,402 | 29 | 24
  pH=7.5; Week 0, n=388,402: number analyzed (Participants) | 388 | 402
  pH=7.5; Week 0, n=388,402 | 13 | 11
  pH=8; Week 0, n=388,402: number analyzed (Participants) | 388 | 402
  pH=8; Week 0, n=388,402 | 6 | 7
  pH=8.5; Week 0, n=388,402: number analyzed (Participants) | 388 | 402
  pH=8.5; Week 0, n=388,402 | 1 | 1
  pH=5; Week 26, n=347,343: number analyzed (Participants) | 347 | 343
  pH=5; Week 26, n=347,343 | 80 | 100
  pH=5.5; Week 26, n=347,343: number analyzed (Participants) | 347 | 343
  pH=5.5; Week 26, n=347,343 | 107 | 104
  pH=6; Week 26, n=347,343: number analyzed (Participants) | 347 | 343
  pH=6; Week 26, n=347,343 | 69 | 70
  pH=6.5; Week 26, n=347,343: number analyzed (Participants) | 347 | 343
  pH=6.5; Week 26, n=347,343 | 42 | 23
  pH=7; Week 26, n=347,343: number analyzed (Participants) | 347 | 343
  pH=7; Week 26, n=347,343 | 19 | 23
  pH=7.5; Week 26, n=347,343: number analyzed (Participants) | 347 | 343
  pH=7.5; Week 26, n=347,343 | 17 | 18
  pH=8; Week 26, n=347,343: number analyzed (Participants) | 347 | 343
  pH=8; Week 26, n=347,343 | 7 | 5
  pH=8.5; Week 26, n=347,343: number analyzed (Participants) | 347 | 343
  pH=8.5; Week 26, n=347,343 | 5 | 0
  pH>9; Week 26, n=347,343: number analyzed (Participants) | 347 | 343
  pH>9; Week 26, n=347,343 | 1 | 0

36. Secondary Outcome: Number of Participants With Different Number of Erythrocytes in Urine at Week 0 and Week 26
Description: Urine samples were collected for analysis of erythrocyte count. Only those participants available at the specified time points were analyzed represented by n=X,X in the category titles. Number of participants with different number of erythrocytes in urine at Week 0 and Week 26 are presented.
Time Frame: Week 0 and Week 26
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 400 | 413
Participants
  None Seen; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  None Seen; Week 0, n=171,187 | 119 | 101
  0 to 1; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  0 to 1; Week 0, n=171,187 | 34 | 51
  1 to 3; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  1 to 3; Week 0, n=171,187 | 9 | 14
  3 to 5; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  3 to 5; Week 0, n=171,187 | 3 | 12
  5 to 10; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  5 to 10; Week 0, n=171,187 | 2 | 4
  10 to 15; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  10 to 15; Week 0, n=171,187 | 0 | 2
  15 to 25; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  15 to 25; Week 0, n=171,187 | 2 | 1
  50 to 100; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  50 to 100; Week 0, n=171,187 | 0 | 1
  >100; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  >100; Week 0, n=171,187 | 2 | 1
  None Seen; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  None Seen; Week 26, n=166,144 | 98 | 79
  0 to 1; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  0 to 1; Week 26, n=166,144 | 48 | 36
  1 to 3; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  1 to 3; Week 26, n=166,144 | 8 | 19
  3 to 5; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  3 to 5; Week 26, n=166,144 | 4 | 3
  5 to 10; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  5 to 10; Week 26, n=166,144 | 4 | 4
  25 to 50; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  25 to 50; Week 26, n=166,144 | 1 | 2
  50 to 100; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  50 to 100; Week 26, n=166,144 | 2 | 0
  >100; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  >100; Week 26, n=166,144 | 1 | 1

37. Secondary Outcome: Number of Participants With Different Number of Leukocytes in Urine at Week 0 and Week 26
Description: Urine samples were collected for analysis of leukocyte count. Only those participants available at the specified time points were analyzed represented by n=X,X in the category titles. Number of participants with different number of leukocytes in urine at Week 0 and Week 26 are presented.
Time Frame: Week 0 and Week 26
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 400 | 413
Participants
  None Seen; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  None Seen; Week 0, n=171,187 | 69 | 67
  0 to 1; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  0 to 1; Week 0, n=171,187 | 27 | 31
  1 to 3; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  1 to 3; Week 0, n=171,187 | 20 | 18
  3 to 5; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  3 to 5; Week 0, n=171,187 | 16 | 13
  5 to 10; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  5 to 10; Week 0, n=171,187 | 17 | 19
  10 to 15; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  10 to 15; Week 0, n=171,187 | 7 | 6
  15 to 25; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  15 to 25; Week 0, n=171,187 | 5 | 11
  25 to 50; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  25 to 50; Week 0, n=171,187 | 5 | 11
  50 to 100; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  50 to 100; Week 0, n=171,187 | 1 | 7
  >100; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  >100; Week 0, n=171,187 | 4 | 3
  Innumerable; Week 0, n=171,187: number analyzed (Participants) | 171 | 187
  Innumerable; Week 0, n=171,187 | 0 | 1
  None Seen; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  None Seen; Week 26, n=166,144 | 65 | 44
  0 to 1; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  0 to 1; Week 26, n=166,144 | 25 | 29
  1 to 3; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  1 to 3; Week 26, n=166,144 | 22 | 20
  3 to 5; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  3 to 5; Week 26, n=166,144 | 10 | 15
  5 to 10; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  5 to 10; Week 26, n=166,144 | 22 | 14
  10 to 15; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  10 to 15; Week 26, n=166,144 | 8 | 5
  15 to 25; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  15 to 25; Week 26, n=166,144 | 3 | 3
  20 to 50; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  20 to 50; Week 26, n=166,144 | 0 | 1
  25 to 50; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  25 to 50; Week 26, n=166,144 | 5 | 6
  50 to 100; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  50 to 100; Week 26, n=166,144 | 5 | 5
  >100; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  >100; Week 26, n=166,144 | 1 | 1
  Innumerable; Week 26, n=166,144: number analyzed (Participants) | 166 | 144
  Innumerable; Week 26, n=166,144 | 0 | 1

38. Secondary Outcome: Change From Baseline in Total Cholesterol (TC), Low-density Lipoprotein Cholesterol (LDL-c), High Density Lipoprotein (HDL-c), Triglycerides (TG) and Free Fatty Acids (FFA) at Week 10 and Week 26
Description: Lipid parameters included TC, LDL-c, HDL-c, TG and FFA. The Baseline value was the last available non-missing value prior to the first dose of the randomized treatment, thus Baseline was Day -1. Change from Baseline is defined as the post-Baseline value minus the Baseline value. LDL-c and FFA were collected as part of the lipid panel and results were reviewed by investigators for individual participants. Change from Baseline at Week 10 and Week 26 was not assessed for these parameters. Analysis of these parameters was not a specific study objective and would not have any impact on study conclusions. Only those parameters with data values have been presented. Only those participants available at the specified time points were analyzed represented by n=X,X in the category titles.
Time Frame: Baseline, Week 10 and Week 26
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per Liters
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 400 | 413
Millimoles per Liters
  TC: Week 10, n=376,393: number analyzed (Participants) | 376 | 393
  TC: Week 10, n=376,393 | -0.244 (0.8047) | 0.041 (0.7425)
  TC: Week 26, n=348,351: number analyzed (Participants) | 348 | 351
  TC: Week 26, n=348,351 | -0.059 (0.8721) | 0.073 (0.8232)
  HDL-c: Week 10, n=376,393: number analyzed (Participants) | 376 | 393
  HDL-c: Week 10, n=376,393 | -0.041 (0.1944) | 0.016 (0.1810)
  HDL-c: Week 26, n=348,351: number analyzed (Participants) | 348 | 351
  HDL-c: Week 26, n=348,351 | -0.013 (0.2102) | 0.005 (0.2138)
  TG: Week 10, n=376,393: number analyzed (Participants) | 376 | 393
  TG: Week 10, n=376,393 | -0.039 (1.3563) | -0.065 (0.8045)
  TG: Week 26, n=348,351: number analyzed (Participants) | 348 | 351
  TG: Week 26, n=348,351 | 0.025 (1.1949) | -0.028 (0.9342)

39. Secondary Outcome: Number of Participants With Vital Signs of Clinical Concern
Description: Vital signs included systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse rate values. Assessment of vitals were performed with the participant in a semi recumbent or seated position having rested in this position for at least 5 minutes before each reading. The potential clinical concern values were: SBP: <100 millimeters of mercury (mmHg) and >170 mmHg, DBP: <50 mmHg and >110 mmHg and pulse rate: <50 beats per minute (bpm) and > 120 bpm. Number of participants with vital signs of clinical concern are presented.
Time Frame: Up to 30 weeks
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 397 | 411
Participants
  SBP: < 100 mmHg | 21 | 20
  SBP: > 170 mmHg | 27 | 30
  DBP: < 50 mmHg | 1 | 4
  DBP: > 110 mmHg | 1 | 5
  Pulse Rate: < 50 bpm | 4 | 9
  Pulse Rate: > 120 bpm | 3 | 1

40. Secondary Outcome: Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) Parameters
Description: A single 12-lead ECG recordings were performed in a participant in semi recumbent position for 10 to 15 minutes before obtaining the ECG. Any clinically significant favorable and unfavorable findings are reported.
Time Frame: Up to 30 weeks
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
Number analyzed (Participants) | 384 | 394
Participants
  Clinically Significant Change: Favorable | 18 | 9
  Clinically Significant Change: Unfavorable | 4 | 5

ADVERSE EVENTS:
Time Frame: Up to 26 weeks
Description: On-treatment SAEs and non-serious AEs were collected for Safety Population which comprised of all participants who receive at least 1 dose of randomized study medication.
Arm/Group | Albiglutide + Insulin Glargine | Insulin Lispro + Insulin Glargine
All-Cause Mortality (participants affected / at risk) | 0/400 | 1/413
Serious Adverse Events (participants affected / at risk) | 23/400 | 31/413
Other Adverse Events (participants affected / at risk) | 114/400 | 101/413
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albiglutide + Insulin Glargine (N=400) | Insulin Lispro + Insulin Glargine (N=413)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2)
Atrial flutter (Cardiac disorders) | 1 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Osteomyelitis (Infections and infestations) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (6)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Perineal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Conductive deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albiglutide + Insulin Glargine (N=400) | Insulin Lispro + Insulin Glargine (N=413)
Influenza (Infections and infestations) | 24 (30) | 36 (42)
Viral upper respiratory tract infection (Infections and infestations) | 25 (33) | 34 (39)
Diarrhoea (Gastrointestinal disorders) | 31 (51) | 18 (19)
Urinary tract infection (Infections and infestations) | 22 (25) | 23 (24)
Nausea (Gastrointestinal disorders) | 37 (53) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-09-24): https://cdn.clinicaltrials.gov/large-docs/27/NCT02229227/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT02229227/SAP_001.pdf